CLINICAL TRIAL: NCT04990583
Title: mHealth Facilitated Intervention to Improve HIV Pre-Exposure Prophylaxis Adherence
Acronym: SMART PrEP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants during COVID-19.
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012820
Record Dates: First submitted 2021-03-08; First posted 2021-08-04 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2020-11

CONDITIONS: Pre-Exposure Prophylaxis; Telemedicine; Medication Adherence
Keywords: PrEP; Adherence; mHealth
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carium Condition (Experimental): Participants assigned to the Carium condition will receive a single session intervention and receive 12 months of access to the Carium adherence application.
  Interventions: Behavioral: Face-to-Face PrEP Adherence Intervention Based on LifeSteps; Behavioral: Adherence Coaching Facilitated by Carium Adherence App
- Control Condition (Active Comparator): Participants assigned to the Control condition will receive a single session intervention only.
  Interventions: Behavioral: Face-to-Face PrEP Adherence Intervention Based on LifeSteps

INTERVENTIONS:
Behavioral: Face-to-Face PrEP Adherence Intervention Based on LifeSteps — This single session intervention, based on LifeSteps, will occur with a study adherence coach either in-person or remotely via HIPAA compliant videoconferencing software. The topics covered during the session will include: experience taking PrEP, risk behavior education, mental health and substance use as barriers to adherence, other barriers to adherence, formulating a dosing schedule, storing and transporting medications, and response to slips in adherence. Participants assigned to the Carium condition will also receive an introduction to the Carium app.
Behavioral: Adherence Coaching Facilitated by Carium Adherence App — The Carium app will be used to deliver medication reminders to participants, track medication adherence, engage in two-way secure messaging with participants, and connect with participants through a secure video feature. The adherence coach will use the secure messaging feature to support the participant with their adherence
  Arms: Carium Condition

SUMMARY:
If taken every day, PrEP is an effective method for preventing HIV. However, many prescribed PrEP in the U.S. do not take it every day, as prescribed. The goal of this study is to develop and test an intervention, facilitated by a mobile app, meant to improve adherence to PrEP. To that end, 60 individuals prescribed PrEP who do not take their PrEP every day as prescribed will be recruited. Participants will complete an initial research interview, receive a one-on-one PrEP adherence session with an adherence coach, and complete follow-up interviews at 1, 3, 6, and 12 months. In addition, some participants will be randomized to receive access to a mobile app and adherence coaching via the app for 12-months. The primary outcome is self-reported adherence to PrEP. This study will examine whether this intervention is effective at improving adherence to PrEP, is feasible to use, and found acceptable by those who use it.

DETAILED DESCRIPTION:
HIV pre-exposure prophylaxis (PrEP), involves the use of antiretroviral (ART) medications (Truvada or Descovy) by persons uninfected with HIV to prevent HIV acquisition. The efficacy of PrEP for preventing HIV acquisition is highly impacted by one's medication adherence. Within the U.S., adherence to PrEP is suboptimal. Commonly cited barriers to PrEP adherence include forgetfulness, low HIV risk perception, stigma, and cost. There is a need for interventions that improve adherence to PrEP, are readily disseminable, and that make efficient use of resources. To that end the current project will examine the feasibility, acceptability, and preliminary efficacy of an intervention tailored for PrEP adherence, facilitated by mHealth. Individuals prescribed PrEP (n = 60) who report taking, on average, fewer than 6 doses per week in the past month will be recruited. Participants will be randomly assigned to the intervention (Carium) or control condition. Data collection will consist of a baseline interview and follow-ups at 1, 3, 6, and 12 months. The primary outcome is PrEP adherence. PrEP adherence will be measured via self-report, pill counts, and use of a urine test developed by UrSure. The urine test is for research use only and will only be used to detect the presence of PrEP in urine if participants self-report taking PrEP in the last 48 hours. It is expected that participants in the Carium condition, relative to control, will report better adherence to PrEP.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* has a prescription for PrEP
* received first prescription for PrEP at least one month ago
* reports taking an average of fewer than 6 PrEP doses per week of over the past month
* has phone that is compatible with the Carium app.

Exclusion Criteria:

* cognitive impairment that would jeopardize informed consent and/or intervention comprehension
* active psychosis
* not fluent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in PrEP Adherence | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  PrEP adherence will be measured via self-report and confirmed by examining concentration of PrEP in participants' urine.

SECONDARY OUTCOMES:
Pill counts | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  Pill counts of PrEP medication will occur in-person or remotely. Date of prescription will be compared to the number of pills remaining.
PrEP Care Retention | 12-month follow-up.
  Medical records will be examined to confirm retention in PrEP care. PrEP care retention will be defined as attending 3-month clinical appointments (+/- 1 month). This information will be extracted from participants' medical records at the 12-month follow-up.
HIV/STI Status | Baseline and 12-month follow-up.
  Results of HIV and STI tests will be extracted from participants' medical records.
Alcohol and Drug Use | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  Daily alcohol and drug use will be assessed with the Timeline Followback (TLFB). The TLFB will provide data on the number of standard drinks consumed per day and types of drug classes used each day.
HIV Risk Behavior | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  The Timeline Followback interview will be used to assess daily drug and sex risk behavior. In addition, the HIV Risk Assessment Battery (RAB) will serve as a measure of overall sex and drug risk.
Center for Epidemiologic Studies Depression Scale (CES-D) | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  The CESD will be used to measure level of depressive symptoms. This measure is widely used and has good sensitivity and specificity and high internal consistency.
PrEP Care Dropout and Non-Adherence | 12-month follow-up.
  Participants who have dropped out of PrEP care or report a period of non-adherence, will be asked open-ended questions at the 12-month follow-up to assess the reasons for treatment dropout and/or non-adherence.
Treatment Received | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  Receipt of case management, psychiatric, substance use, and other treatment services will be assessed with the Treatment Services Review.
Medications | Baseline, 1-, 3-, 6-, and 12-month follow-ups.
  Participants will also be asked about their use of medications for medical, psychiatric, or substance use indications.

OTHER OUTCOMES:
Indices of Feasibility | 12-month follow-up.
  Patient eligibility rate, enrollment refusal rate, rate of recruitment, and follow-up completion rate in order to evaluate the feasibility of conducting a subsequent larger study using this protocol.
Indices of Acceptability | 12-month follow-up.
  The study team will compile a study dropout rate and intervention session completion rate, as indices of acceptability.
System Usability Scale | 6- and 12-month follow-up.
  Satisfaction with the intervention will be assessed with the System Usability Scale.
Paradata from Carium App | 12-month follow-up
  Paradata will be extracted from the Carium app. This information will provide context about how often participants used the app in the intervention condition.
Intervention Feedback | 12-month follow-up.
  A semi-structured interview will be conducted with participants. The point of the semi-structured interview will be to get feedback about the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States